CLINICAL TRIAL: NCT05962541
Title: Non-inferiority, Phase IV, Open-label, Randomized Controlled Trial of Vesical Imaging- Reporting and Data System (VI-RADS) Followed by Primary Photodynamic Trans-urethral Resection of Bladder Tumours (PDD-TURBT) Versus Conventional White-light TURBT Plus Repeated-TURBT (Re-TURBT) in Non-Muscle Invasive Bladder Cancers (NMIBCs) Candidate for Second Look and Resection
Brief Title: Vesical Imaging-Reporting and Data System (VI-RADS) Followed by Photodynamic Trans-urethral Resection of Bladder Tumours (PDD-TURBT) to Avoid Secondary Resections (Re-TURBT) in Non-Muscle Invasive Bladder Cancers (NMIBCs)
Acronym: CUT-less
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Del Giudice, Chief Investigator, MD, PhD, Assistant Professor, Consultant Urologic Surgeon, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N764J-20022023
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Non-muscle-invasive Bladder Cancer; Non-Muscle Invasive Bladder Urothelial Carcinoma; High Risk Non-Muscle Invasive Bladder Urothelial Carcinoma
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Intervention Model Description: Italian, single-center, phase IV, open-label, randomized controlled trial, with patients randomized in a 1:1 ratio to one of two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPD-TURBT (no Re-TURBT) (Experimental): Primary PDD-TURBT, not followed by Re-TURBT
  Interventions: Drug: PDD-TURBT with hexaminolevulinate (Hexvix®); Device: Power Led Saphira (TM)
- WL TURBT plus Re-TURBT (Standard of Care) (No Intervention): Standard of care consisting in primary WL TURBT followed by WL Re-TURBT within 2 - 6 weeks from initial WL TURBT

INTERVENTIONS:
Drug: PDD-TURBT with hexaminolevulinate (Hexvix®) — In order to undergo PDD-TURBT, all eligible patients in the experimental arm will be administered the photosensitizer hexaminolevulinate (85 mg in 50 ml of phosphate buffered saline, Hexvix®) on an inpatient setting through a urethral catheterization of the participant's bladder. During the PDD-TURBT surgery, the bladder will be illuminated with blue light (wavelength 380-450 nm). The operating rooms of the participant institutions will therefore need to have the specialized equipment consisting in the blue-light source (POWER LED SAPHIRA [TM]).
  Other Names: Hexvix®
  Arms: PPD-TURBT (no Re-TURBT)
Device: Power Led Saphira (TM) — This is a light source based on LED technology. It can be used for both White Light (WL) and fluorescence applications in blue light (i.e., Photodynamic diagnosis PDD) for visualizing tumor lesions during trans-urethral resection of bladder tumors (PPD- TURBT).
  Arms: PPD-TURBT (no Re-TURBT)

SUMMARY:
Background: In European Association of Urology (EAU) Guidelines, the vast majority of non-muscle-invasive bladder cancers (NMIBCs) undergo a primary transurethral resection of the bladder tumor (TURBT) followed by a repeat TURBT (Re-TURBT). The Re-TURBT is recommended due to the possibility of residual bladder cancer but is unnecessary in many cases by constituting overtreatment. Currently, no diagnostic strategy or predictive tools have been implemented to further stratify who does or does not benefit from Re-TURBT. Recently, an MRI-based Vesical Imaging Reporting and Data System (VI-RADS) score has been developed to stage as to the preoperative probability of muscle invasion, which could potentially exclude those who do not require a Re-TURBT when a primary high-quality resection is delivered. As such, performing TURBT with standard white light (WL) cystoscopy is known to miss many bladder tumours, which may be poorly visible, and a technique known as with photodynamic diagnosis (PDD) results in lower residual tumor and lower early intravesical recurrence rates. PDD is performed using violet light to improve the detection of these lesions not easily visible with WL cystoscopy.

Methods/Aims: The investigators propose an Italian, single-center, phase IV, open-label, non-inferiority, randomized controlled trial, in which participants (n=112) who had already received a mpMRI/VI-RADS score, are randomized to receive PDD-TURBT, no Re-TURBT versus standard of care represented by conventional WL-TURBT followed by WL-Re-TURBT. The primary outcome is proportions of early recurrence in the urinary bladder. Secondary outcomes will include proportions of late BCa recurrence, late disease-free interval, time to progression to MIBC, patient's quality of life assessment, and cost-analysis.

Perspective: The CUT-less trial aims to respond to this unmet need through a non-inferiority randomized clinical study potentially shaping the perspective for a paradigm shift towards a more personalized, socially, and economically sustainable updated NMIBC therapeutic pathway.

Implications: The current clinical trial proposal is aiming to achieve a paradigm shift in the oncological and socio-economical management of urothelial malignancies of the urinary bladder. Our first concern is indeed to guarantee a safe and ground-breaking strategy to manage the pathway of such patients in order to guarantee the non-inferior oncologic safety (and possibly superiority) when compared to the current standard of care.

Additionally, if our hypotheses are confirmed, the investigators will be able to significantly relieve these patients from the oncologic burden of an already invasive and arduous bladder cancer care path. Finally, safely avoiding an unnecessary, expensive surgical procedure will bring significant social and economic benefits to the EU healthcare system and possibly worldwide.

DETAILED DESCRIPTION:
BACKGROUND, STATE OF THE ART and RATIONALE FOR THE INTERVENTIONS

The vast majority (75-80%) of bladder cancers (BCa) patients present with disease confined either to the mucosa (stage Ta, carcinoma in situ [CIS]) or the submucosa (stage T1) according to the tumor, node, and metastasis (TNM) classification system. These tumours that do not invade the detrusor muscle of the urinary bladder are defined as superficial, non-invasive, or non-muscle invasive bladder cancers (NMIBC) to differentiate them from the less common, but significantly more deadly muscle invasive bladder cancers (MIBC; stage T2 - T4).

Although the initial procedure for surgical management of both NMIBC and MIBC tumours is a trans-urethral resection of bladder tumor (TURBT), it serves different purposes for NMIBC when compared with MIBC. For NMIBC, TURBT acts as both a diagnostic and a therapeutic procedure, but for MIBC patients, TURBT is only a diagnostic procedure, as additional radical intervention, such as radical cystectomy (RC), are usually required.

However, there are many potential issues that can affect TURBT performance, including a high degree of operator dependence for optimal outcomes. Along these lines, one particular issue is that many of the so-called early BCa recurrences are actually incomplete resections during initial TURBT. Incomplete resections can lead also to understaging (i.e., inaccurate discrimination between NMIBC and MIBC), which can adversely affect the survival of the patient. Incomplete tumor resection and residual tumor rates vary between 33% and 76% for all cases, with rates of 27-72% and 33-78% for Ta and T1 tumours, respectively. Also, underestimation of tumor depth invasion at first TURBT has been demonstrated in up to 7-30% of cases, increasing up to 45-51% in those with T1 tumours where no detrusor muscle was sampled in the specimen after initial TURBT.

Based on these above issues, European Association of Urology (EAU) Guidelines recommend a second look and resection (i.e., re-do TURBT [Re-TURBT]) 2 to 6 weeks following the primary TURBT in cases of (I) incomplete initial TURBT or doubt about completeness of a TURBT, (II) if there is no detrusor muscle in the specimen after initial TURBT, and (III) in all T1 tumours.

As such, if Re-TURBT is to be considered an "emergency rescue" performed because of the suboptimal quality of the initial TURBT, this can result in significant detriments to the patient's quality of life (QoL) (e.g., second hospitalization, second anesthesia, potential risk for complications, delay in definitive treatment etc.). These can result in additional negative social implications (e.g., productivity loss, indirect costs etc.) and health-care-related costs (e.g., surgical procedure costs, in-hospital recovery costs, postoperative care etc.).

The CUT-less study aims to address these major oncological, economic, and social unmet needs related to the current EAU BCa algorithm throughout a phase IV, open-label, non-inferiority randomized controlled trial. In particular, one of our aims is trying to avoid unnecessary Re-TURBT by utilizing intraoperative visually enhanced photodynamic assisted TURBT (PDD-TURBT) among those who had already been evaluated by multiparametric magnetic resonance (mpMR) image-based staging before the initial TURBT as a combined novel strategy. In doing so, the investigators hope to select for those in whom a Re-TURBT would normally be recommended, unnecessarily. The investigators will compare this cohort to one that follows the current standard of care algorithm, (i.e., conventional white light [WL] initial TURBT followed by WL-Re-TURBT). The investigators will examine the relative proportions of early BCa recurrence within the first 4.5 months after randomization. This would be the time between randomization, surgical TURBTs (i.e., 1.5 months) and first follow-up cystoscopy which is set at 3 months according to the International NMIBC Clinical trial Guidelines.

The primary objectives of the CUT-less trial are indeed to provide the highest level of evidence demonstrating non-inferiority between of this novel multidisciplinary and translational approach integrating functional MRI and intraoperative visually assisted enhanced trans-urethral surgery and the current EAU BCa pathway. This will potentially lead to the redefinition of the criteria for Re-TURBT selection and will avoid unnecessary surgical procedures in up to half of diagnosed NMIBCs. The impact of such paradigm shift will transform the patient's perspective in their own BCa care and will limit the social and economic burden of BCa management across the EU and hopefully worldwide.

STUDY AIMS, DESIGN and METHODOLOGICAL FRAMEWORK

Overall aim To utilize our expertise in mpMRI of the bladder diagnostics for pre-TURBT staging purposes, intraoperative TURBT optical imaging enhancement by PDD-guided primary resection in order to potentially shift clinical practice. In doing so, the investigators seek to improve the therapeutic algorithm and personalization for NMIBC treatment by not performing those Re-TURBT procedures which could be safely omitted.

Sample Size Calculation The cohort of interest will be represented by intermediate/high-risk NMIBCs who are currently those eligible for Re-TURBT according to EUA Guidelines. For the primary outcome of the proportion of early BCa recurrence (i.e., within 4.5 months follow-up) between the two arms, the investigators acknowledge that rates of early BCa recurrence detection among NMIBCs undergoing TURBT along with adjuvant intravesical BCG immunotherapy in a population, with equally distributed literature-defined risk factors for BCa recurrences, have been shown to be 10% according to available literature.

For the non-inferiority hypothesis, using 80% power and a 5% one sided-alpha, using an estimate for detection rate of early BCa recurrence among intermediate/high-risk NMIBCs of 7.5% and using a margin of clinical unimportance of 10%, n=112 patients per arm will be required. The choice of 10% as the margin of non-inferiority represents a difference that would be considered clinically unimportant in the detection rate for the event of early BCa recurrence in a population already screened by mpMRI and VI-RADS score determination for the risk of disease understaging.

To achieve this, prior to randomization, the investigators will screen potential eligible participants by VI-RADS score determination and will exclude patients suspected for MIBC (15-20%) and, from the remaining NMIBCs, exclude low risk disease (25-30%). Furthermore, the investigators predict 35-40% of these patients will be recruited based on willingness to participate or missed opportunities for recruitment.

Thus, total subjects required in study would be n=284. Accounting for 15% withdrawal/loss to follow up, n=327 men will need to be recruited.

GROUND-BREAKING AMBITION OF THE PROPOSAL AND ADVANCEMENT OF KNOWLEDGE OVER THE STATE OF THE ART

BCa is a high priority area for research into both clinical and cost-effective management and the findings from the CUT-less trial will be relevant and important to patient needs over the next years across the EU and worldwide.

TURBT is the standard of care both to diagnose and treat the vast majority of NMIBCs. Nonetheless, to overcome the intrinsic limitations of TURBT, to achieve the desired complete resection, and to correct potential staging errors, a second endoscopic procedure (i.e., Re-TURBT) is recommended by EUA Guidelines for most intermediate and high-risk NMIBCs categories. However, there is still no currently available strategy to select the ideal candidate for this.

Notably, from a patient perspective, there are often considerable anxieties about transurethral resection procedures, risk of recurrences, and progression requiring additional therapies with potential mortality and long-term morbidity. TURBTs in general, are associated with possible significant postoperative and long-term complications and morbidity ranging from 5.1% to 43.3% according to the different series. Specifically, the potential for complications during Re-TURBT is not trivial and hemorrhage, the need for blood transfusion, or bladder perforation can negatively impact patient care and lead to delays in treatment, ultimately influencing survival outcomes. Any TUR itself is therefore associated with reduced QoL, including in both mental and physical health domains. Substantial reductions in health related QoL are most likely to come from repeated hospitalizations, surgical complications, invasive adjuvant intravesical treatments, and radical or palliative treatments for progression. As consequence, a secondary resection performed 2 to 6 weeks from the primary resection represents an additional burden in an already arduous BCa pathway. To our knowledge this surgical scenario has never been scrutinized in the framework of a RCT despite the lack of evidence to uniformly support Re-TURBT in every case. Moreover, both European and American series had reported that performing Re-TURBT did not impact long-term progression-free survival and that the tumor status at repeat TUR had only a marginal role in influencing long-term cancer-specific survival.

Additionally, NMIBC is one of the most expensive cancers to manage on a per patient basis because of its high prevalence, high recurrence rate, need for adjuvant treatments, and the requirement for long-term surveillance protocols. Because of the protracted clinical course of early-stage disease, its prevalence relative to MIBC, and its procedure-oriented surveillance, the associated cumulative medical payments are generally more substantial than those for advanced disease. The average per capita spending for NMIBC is increasing in the last two decades, from €7000 to €9000. These increasing costs are mainly attributable to the more frequent use of endoscopy (e.g., cystoscopy, TURBT, Re-TURBT) and the adjuvant intravesical therapies. TURBT accounts for a substantial portion of total bladder treatment costs ranging from €3000 to €6000 depending on whether patients are discharged following the procedure or admitted for inpatient care.

Given these urgent needs for optimizing the NMIBC algorithm, the CUT-less trial will explore a novel multidisciplinary approach for minimizing the burden of surgical exposure to patients and for resizing the costs to the EU health care systems by redefining the selection criteria for NMIBC candidates for Re-TURBT procedures.

In conclusion, the currently available EAU Guidelines rely on conflicting and out of date evidence which do not offer a contemporary viewpoint as to the role of Re-TURBT. Our updated protocol which utilizes both mpMRI diagnostic imaging and PDD guided resections will be closely examined in the CUT-less trial, with goal of more personalized, both socially and economically sustainable updated NMIBC therapeutic pathways for use in the EU.

ELIGIBILITY:
Inclusion Criteria:

1. Female and Male patients at least 18 years old referred for clinical suspicion of primary or recurrent BCa who have been advised to undergo TURBT.
2. Patients with a TUR-confirmed diagnosis of NMIBC and candidate for second look and resection (Re-TURBT) according to EAU Guidelines [6].
3. No imaging evidence (i.e., mpMRI/VI-RADS score 1 or 2) of muscle-invasive, locally advanced, or metastatic BCa (i.e., only confirmed CIS, Ta, T1, N0, M0 will be considered eligible).
4. Patients who did or did not receive previous BCG immunotherapy (i.e., BCG naïve and non-naïve patients).
5. Fit to undergo all procedures listed in protocol.
6. Able to provide written informed consent.

Exclusion Criteria:

1. Contraindication to TURBT and/or Re-TURBT.
2. Initial TURBT diagnosis of MIBC (i.e., T2) or locally advanced BCa (i.e., T3-T4).
3. Preoperative evidence of metastatic disease (i.e., cN1 - N3 and/or cM1).
4. Visual evidence of low-risk NMIBC (solitary tumor, < 1 cm) before initial TURBT.
5. Visual evidence of MIBC on preliminary cystoscopy (i.e., non-papillary or sessile mass attached directly by its base without a stalk).
6. TURBT diagnosis of NMIBCs not eligible for Re-TURBT according to EAU Guidelines (i.e., Ta-LG; Ta-HG with detrusor muscle in the specimen; primary CIS) [6].
7. Concomitant Upper tract (kidney or ureteric) tumours on imaging.
8. Contraindication to adjuvant intravesical BCG immunotherapy.
9. Unfit to undergo any procedures listed in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of EARLY Bladder Cancer (BCa) recurrences | within 4.5 months following primary intervention
  The proportion of early BCa recurrences (i.e., within 4.5 months follow-up) in those non-muscle invasive bladder cancer (NMIBC) treated by standard of care (i.e., TURBT followed by Re-TURBT) compared to our novel algorithm proposal (i.e., primary PDD-TURBT followed by no Re-TURBT).

SECONDARY OUTCOMES:
Proportion of LATE BCa recurrences | after 4.5 months following primary intervention
  To determine the proportion of BCa late recurrences (i.e., after 4.5 months follow-up) in patients with NMIBC treated by standard of care compared to our novel algorithm proposal
Proportion of progression from NMIBC to MIBC | over 3 years follow-up
  To determine the proportion of progression from NMIBC to MIBC in patients with NMIBC treated by standard of care compared to our novel algorithm proposal.
Changes in health-related quality of life (HRQoL) | over 3 years follow-up
  To determine changes in health-related quality of life (HRQoL) resulting from the physical and psychological benefit together with any harms associated with each strategy and with subsequent additional interventions. We will use generic QoL for cost-effectiveness analysis (i.e., EuroQoL Group [EQ]-5D-3L).
Changes in health-related quality of life (HRQoL) | over 3 years follow-up
  To determine changes in health-related quality of life (HRQoL) resulting from the physical and psychological benefit together with any harms associated with each strategy and with subsequent additional interventions. We will use and specific validated questionnaires to assess the outcomes of interest in the NMIBC population (i.e., European Organisation for Research and Treatment of Cancer [EORTC]-QLQ-C30).
Changes in health-related quality of life (HRQoL) | over 3 years follow-up
  To determine changes in health-related quality of life (HRQoL) resulting from the physical and psychological benefit together with any harms associated with each strategy and with subsequent additional interventions. We will use and specific validated questionnaires to assess the outcomes of interest in the NMIBC population (i.e., European Organisation for Research and Treatment of Cancer [EORTC] QLQ-NMIBC24).
Cost-effectiveness analysis | over 3 years follow-up
  To perform a within-trial cost-effectiveness analysis to calculate incremental cost per Re-TURBT avoided and the cost-utility of the experimental approach as measured by the incremental cost per quality-adjusted life year (QALY) gained at 2 years and over patients' lifetime.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico Umberto I Hospital, UOC Urologia SMUC05, Rome, Italy, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein JI, Amin MB, Reuter VR, Mostofi FK. The World Health Organization/International Society of Urological Pathology consensus classification of urothelial (transitional cell) neoplasms of the urinary bladder. Bladder Consensus Conference Committee. Am J Surg Pathol. 1998 Dec;22(12):1435-48. doi: 10.1097/00000478-199812000-00001. PMID 9850170
- [Background] Mariappan P, Zachou A, Grigor KM; Edinburgh Uro-Oncology Group. Detrusor muscle in the first, apparently complete transurethral resection of bladder tumour specimen is a surrogate marker of resection quality, predicts risk of early recurrence, and is dependent on operator experience. Eur Urol. 2010 May;57(5):843-9. doi: 10.1016/j.eururo.2009.05.047. Epub 2009 Jun 6. PMID 19524354
- [Background] Brausi M, Collette L, Kurth K, van der Meijden AP, Oosterlinck W, Witjes JA, Newling D, Bouffioux C, Sylvester RJ; EORTC Genito-Urinary Tract Cancer Collaborative Group. Variability in the recurrence rate at first follow-up cystoscopy after TUR in stage Ta T1 transitional cell carcinoma of the bladder: a combined analysis of seven EORTC studies. Eur Urol. 2002 May;41(5):523-31. doi: 10.1016/s0302-2838(02)00068-4. PMID 12074794
- [Background] Cumberbatch MGK, Foerster B, Catto JWF, Kamat AM, Kassouf W, Jubber I, Shariat SF, Sylvester RJ, Gontero P. Repeat Transurethral Resection in Non-muscle-invasive Bladder Cancer: A Systematic Review. Eur Urol. 2018 Jun;73(6):925-933. doi: 10.1016/j.eururo.2018.02.014. Epub 2018 Mar 6. PMID 29523366
- [Background] Naselli A, Hurle R, Paparella S, Buffi NM, Lughezzani G, Lista G, Casale P, Saita A, Lazzeri M, Guazzoni G. Role of Restaging Transurethral Resection for T1 Non-muscle invasive Bladder Cancer: A Systematic Review and Meta-analysis. Eur Urol Focus. 2018 Jul;4(4):558-567. doi: 10.1016/j.euf.2016.12.011. Epub 2017 Jan 13. PMID 28753839
- [Background] Shindo T, Masumori N, Kitamura H, Tanaka T, Fukuta F, Hasegawa T, Yanase M, Miyake M, Miyao N, Takahashi A, Matsukawa M, Taguchi K, Shigyo M, Kunishima Y, Tachiki H, Tsukamoto T. Clinical significance of definite muscle layer in TUR specimen for evaluating progression rate in T1G3 bladder cancer: multicenter retrospective study by the Sapporo Medical University Urologic Oncology Consortium (SUOC). World J Urol. 2014 Oct;32(5):1281-5. doi: 10.1007/s00345-013-1205-1. Epub 2013 Nov 5. PMID 24190368
- [Background] Kamat AM, Sylvester RJ, Bohle A, Palou J, Lamm DL, Brausi M, Soloway M, Persad R, Buckley R, Colombel M, Witjes JA. Definitions, End Points, and Clinical Trial Designs for Non-Muscle-Invasive Bladder Cancer: Recommendations From the International Bladder Cancer Group. J Clin Oncol. 2016 Jun 1;34(16):1935-44. doi: 10.1200/JCO.2015.64.4070. Epub 2016 Jan 25. PMID 26811532
- [Background] Kobayashi K, Matsuyama H, Kawai T, Ikeda A, Miyake M, Nishimoto K, Matsushita Y, Komura K, Abe T, Kume H, Nishiyama H, Fujimoto K, Oyama M, Miyake H, Inoue K, Mitsui T, Kawakita M, Ohyama C, Mizokami A, Kuroiwa H. Bladder cancer prospective cohort study on high-risk non-muscle invasive bladder cancer after photodynamic diagnosis-assisted transurethral resection of the bladder tumor (BRIGHT study). Int J Urol. 2022 Jul;29(7):632-638. doi: 10.1111/iju.14854. Epub 2022 Mar 15. PMID 35293022
- [Background] Cambier S, Sylvester RJ, Collette L, Gontero P, Brausi MA, van Andel G, Kirkels WJ, Silva FC, Oosterlinck W, Prescott S, Kirkali Z, Powell PH, de Reijke TM, Turkeri L, Collette S, Oddens J. EORTC Nomograms and Risk Groups for Predicting Recurrence, Progression, and Disease-specific and Overall Survival in Non-Muscle-invasive Stage Ta-T1 Urothelial Bladder Cancer Patients Treated with 1-3 Years of Maintenance Bacillus Calmette-Guerin. Eur Urol. 2016 Jan;69(1):60-9. doi: 10.1016/j.eururo.2015.06.045. Epub 2015 Jul 23. PMID 26210894
- [Background] Oddens J, Brausi M, Sylvester R, Bono A, van de Beek C, van Andel G, Gontero P, Hoeltl W, Turkeri L, Marreaud S, Collette S, Oosterlinck W. Final results of an EORTC-GU cancers group randomized study of maintenance bacillus Calmette-Guerin in intermediate- and high-risk Ta, T1 papillary carcinoma of the urinary bladder: one-third dose versus full dose and 1 year versus 3 years of maintenance. Eur Urol. 2013 Mar;63(3):462-72. doi: 10.1016/j.eururo.2012.10.039. Epub 2012 Nov 2. PMID 23141049
- [Background] Waldbillig F, Nientiedt M, Kowalewski KF, Grune B, von Hardenberg J, Nuhn P, Michel MS, Kriegmair MC. The Comprehensive Complication Index for Advanced Monitoring of Complications Following Endoscopic Surgery of the Lower Urinary Tract. J Endourol. 2021 Apr;35(4):490-496. doi: 10.1089/end.2020.0825. Epub 2021 Jan 25. PMID 33222525
- [Background] Nieder AM, Meinbach DS, Kim SS, Soloway MS. Transurethral bladder tumor resection: intraoperative and postoperative complications in a residency setting. J Urol. 2005 Dec;174(6):2307-9. doi: 10.1097/01.ju.0000181797.19395.03. PMID 16280830
- [Background] Angulo JC, Palou J, Garcia-Tello A, de Fata FR, Rodriguez O, Villavicencio H. Second transurethral resection and prognosis of high-grade non-muscle invasive bladder cancer in patients not receiving bacillus Calmette-Guerin. Actas Urol Esp. 2014 Apr;38(3):164-71. doi: 10.1016/j.acuro.2014.01.001. Epub 2014 Mar 7. English, Spanish. PMID 24613147
- [Background] Hemdan T, Johansson R, Jahnson S, Hellstrom P, Tasdemir I, Malmstrom PU; Members of the Urothelial Cancer Group of the Nordic Association of Urology. 5-Year outcome of a randomized prospective study comparing bacillus Calmette-Guerin with epirubicin and interferon-alpha2b in patients with T1 bladder cancer. J Urol. 2014 May;191(5):1244-9. doi: 10.1016/j.juro.2013.11.005. Epub 2013 Nov 11. PMID 24231843
- [Background] Gontero P, Sylvester R, Pisano F, Joniau S, Oderda M, Serretta V, Larre S, Di Stasi S, Van Rhijn B, Witjes AJ, Grotenhuis AJ, Colombo R, Briganti A, Babjuk M, Soukup V, Malmstrom PU, Irani J, Malats N, Baniel J, Mano R, Cai T, Cha EK, Ardelt P, Vakarakis J, Bartoletti R, Dalbagni G, Shariat SF, Xylinas E, Karnes RJ, Palou J. The impact of re-transurethral resection on clinical outcomes in a large multicentre cohort of patients with T1 high-grade/Grade 3 bladder cancer treated with bacille Calmette-Guerin. BJU Int. 2016 Jul;118(1):44-52. doi: 10.1111/bju.13354. Epub 2015 Nov 6. PMID 26469362
- [Background] Svatek RS, Hollenbeck BK, Holmang S, Lee R, Kim SP, Stenzl A, Lotan Y. The economics of bladder cancer: costs and considerations of caring for this disease. Eur Urol. 2014 Aug;66(2):253-62. doi: 10.1016/j.eururo.2014.01.006. Epub 2014 Jan 21. PMID 24472711
- [Background] Leal J, Luengo-Fernandez R, Sullivan R, Witjes JA. Economic Burden of Bladder Cancer Across the European Union. Eur Urol. 2016 Mar;69(3):438-47. doi: 10.1016/j.eururo.2015.10.024. Epub 2015 Oct 25. PMID 26508308
- [Background] Strope SA, Ye Z, Hollingsworth JM, Hollenbeck BK. Patterns of care for early stage bladder cancer. Cancer. 2010 Jun 1;116(11):2604-11. doi: 10.1002/cncr.25007. PMID 20310051
- [Background] Skolarus TA, Ye Z, Zhang S, Hollenbeck BK. Regional differences in early stage bladder cancer care and outcomes. Urology. 2010 Aug;76(2):391-6. doi: 10.1016/j.urology.2009.12.079. Epub 2010 Apr 14. PMID 20394976
- [Background] Babjuk M, Burger M, Capoun O, Cohen D, Comperat EM, Dominguez Escrig JL, Gontero P, Liedberg F, Masson-Lecomte A, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Seisen T, Soukup V, Sylvester RJ. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (Ta, T1, and Carcinoma in Situ). Eur Urol. 2022 Jan;81(1):75-94. doi: 10.1016/j.eururo.2021.08.010. Epub 2021 Sep 10. PMID 34511303
- [Derived] Del Giudice F, Vestri A, Fegatelli DA, Husch T, Belsey J, Nair R, Skinner EC, Chung BI, Pecoraro M, Sciarra A, Franco G, Pradere B, Gazzaniga P, Magloicca FM, Panebianco V, De Berardinis E. VI-RADS followed by Photodynamic Transurethral Resection of Non-Muscle-Invasive Bladder Cancer vs White-Light Conventional and Second-resection: the 'CUT-less' Randomised Trial Protocol. BJU Int. 2025 Feb;135(2):346-354. doi: 10.1111/bju.16531. Epub 2024 Oct 13. PMID 39397266